CLINICAL TRIAL: NCT05222646
Title: Metoclopramide Versus Hyoscine Butylbromide in Shortening Duration of the First Stage of Labor Among Nulliparous Women in Abakaliki
Brief Title: Metoclopramide Versus Hyoscine Butylbromide in Shortening Duration of First Stage of Labour
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uwakwe Emmanuel Chijioke (Other)
Responsible Party: Sponsor-Investigator, Uwakwe Emmanuel Chijioke, Principal Investigator, Alex Ekwueme Federal University Teaching Hospital
Organization: Alex Ekwueme Federal University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AEFUTHA/16/07/2020.4/11/2020
Record Dates: First submitted 2021-10-05; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Duration of Labour
MeSH Terms: interventions — Metoclopramide

STUDY DESIGN:
Intervention Model Description: Will receive single dose of 10mg of Metoclopramide intramuscularly
Who Masked: Participant, Investigator
Masking Description: Will receive 20 mg of Hyoscine bromide,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metoclopramide group (Active Comparator): They will be receiving10mg of Metoclopramide intramuscularly
  Interventions: Drug: Metoclopramide
- Hyoscine bromide group (Active Comparator): They will be receiving 20 mg of Hyoscine bromide
  Interventions: Drug: Metoclopramide

INTERVENTIONS:
Drug: Metoclopramide — Will receive single dose of 10mg of Metoclopramide intramuscularly
  Other Names: Placebo

SUMMARY:
BACKGROUND Prolonged labour can lead to increased maternal and neonatal mortality and morbidity. The risk for complications of prolonged labour is more in poor resource settings. Active management of labour has been shown to decrease the occurrence of prolonged labour. Administering antispasmodics during labour could also lead to faster and more effective dilatation of the cervix. As the evidence to support this is still largely anecdotal around the world, there is a need to conduct clinical trials so as to obtain a valid answer.

DETAILED DESCRIPTION:
BACKGROUND Prolonged labour can lead to increased maternal and neonatal mortality and morbidity. The risk for complications of prolonged labour is more in poor resource settings. Active management of labour has been shown to decrease the occurrence of prolonged labour. Administering antispasmodics during labour could also lead to faster and more effective dilatation of the cervix. As the evidence to support this is still largely anecdotal around the world, there is a need to conduct clinical trials so as to obtain a valid answer.

OBJECTIVE This study is designed to compare the effectiveness of metoclopramide versus hyoscine butyl bromide in shortening the duration of the first stage of labour in Abakaliki.

Methods: This would be an equivalence randomized, double-blinded, placebo-controlled trial among nulliparous women in labour Abakaliki to determine the effectiveness of intramuscular Metoclopramide versus intramuscular Hyoscine bromide in shortening the duration of the first stage of labour. One arm will receive a single dose of 10mg of Metoclopramide intramuscularly, another will receive 20 mg of Hyoscine bromide, the third am will receive 1 ml of sterile water(placebo) intramuscularly. The data obtained will be analysed using Statistical Package for Social Science (IBM SPSS) software (version 20, Chicago II, USA) and the intention to treat the concept. Continuous variables would be presented as mean and standard deviation (Mean ± 2SD), while categorical variables would be presented as numbers and percentages. Logistic regression will also be applied where applicable. A difference with a P-value of ≤ 0.05 will be taken to be statistically significant.

Results: The results will be presented in tables from where conclusions will be drawn

CONCLUSION KEYWORD Prolonged labour, Metoclopramide, Hyoscine Bromide, the active phase of labour

ELIGIBILITY:
Inclusion Criteria:

1. All nullipara who gave consent

Exclusion Criteria:

1. those who refused consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-08-03 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Duration of first stage of labour | 6 months
  Duration of first stage of labour

CONTACTS AND LOCATIONS:
Overall Officials: Uwakwe DR Emmanuel Chijioke, PART 1, Principal Investigator — Alex Ekwueme Federal University Teaching Hospital
Locations (1):
- AEFUTHA, Abakaliki, Ebonyi State, Nigeria